CLINICAL TRIAL: NCT00790816
Title: An Open-Label Phase Ib Continuation Study of Lapatinib Monotherapy or Lapatinib in Combination With Other Anti-Cancer Treatment in Patients With Solid Tumors
Brief Title: Continuation Study of Lapatinib Monotherapy or Lapatinib in Combination With Other Anti-cancer Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111767
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Neoplasms, Breast
Keywords: Cancer; lapatinib; Combination therapy; Chronic administration
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Study Drug
  Interventions: Drug: Lapatinib; Drug: Lapatinib in combination with an anti-cancer agent as specified by parent protocol
- Group 2 (Experimental): Study Drug
  Interventions: Drug: Lapatinib in combination with an anti-cancer agent; Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib in combination with an anti-cancer agent — Lapatinib in combination with paclitaxel, letrozole, capecitabine, capecitabine/oxaliplatin, gemcitabine, docetaxel, trastuzumab, FOLFOX4, or FOLFIRI
  Arms: Group 2
Drug: Lapatinib — Lapatinib monotherapy
Drug: Lapatinib in combination with an anti-cancer agent as specified by parent protocol — Lapatinib in combination with an anti-cancer agent as specified by parent protocol
  Arms: Group 1

SUMMARY:
This study is designed to provide continued access to lapatinib as monotherapy or as part of a combination regimen to cancer subjects who are currently participating in a phase I trial that has met its study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a Phase I lapatinib trial that has met its study objectives.
* Ability to understand and provide written informed consent to participate in this study.
* Male or female greater than or equal to 18 years of age.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods stated in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least two to four weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential, has a negative serum pregnancy test at baseline, and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception from two weeks prior to the administration of study drug and throughout the entire active study treatment period until four weeks after the last dose of study medication.

Exclusion Criteria:

* Permanent discontinuation of lapatinib in the previous study due to intolerance or treatment failure.
* Is a pregnant or lactating female.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or baseline investigations.
* Currently receiving treatment with any medications listed on the prohibited medication listed in the protocol
* Has Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Have current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-10; Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Initiation of study treatment to discontinuation of study treatment

SECONDARY OUTCOMES:
Efficacy | Initiation of study treatment to discontinuation of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (15):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Salt Lake City, Utah
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Amsterdam, Netherlands
- South Korea (2):
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Songpa-gu, Seoul
- Novartis Investigative Site, Hospitalet de Llobregat (Barcelona), Spain